CLINICAL TRIAL: NCT00838084
Title: Single-Ascending Dose, Safety, Tolerability, Pharmacokinetic, and Pharmacodynamic Study of LY2811376 in Healthy Subjects
Brief Title: A Safety Study of LY2811376 Single Doses in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 12852; I3J-MC-LACE
Record Dates: First submitted 2009-01-23; First posted 2009-02-06 (Estimated); Last update posted 2009-07-15 (Estimated); Status verified 2009-07

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — LY2811376

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- LY2811376 Part 1 (Experimental): LY2811376 (5 mg up to 500 mg); once a day or twice a day for 1 day in up to 3 periods.
  Interventions: Drug: LY2811376
- Placebo Part 1 (Placebo Comparator): once a day or twice a day for 1 day in up to 3 periods.
  Interventions: Drug: Placebo
- LY2811376 - Part 2 low dose (Experimental): Single dose of LY2811376, dose determined by part 1
  Interventions: Drug: LY2811376
- LY2811376 - Part 2 high dose (Experimental): Single dose of LY2811376, dose determined by part 1
  Interventions: Drug: LY2811376
- Placebo Part 2 (Placebo Comparator): single dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY2811376 — Oral capsules
  Arms: LY2811376 - Part 2 high dose; LY2811376 - Part 2 low dose; LY2811376 Part 1
Drug: Placebo — Oral capsules
  Arms: Placebo Part 1; Placebo Part 2

SUMMARY:
This is a Phase 1 study in healthy subjects to evaluate the safety and tolerability of LY2811376 single doses, how the body handles the drug, and the drug's effect on the body.

DETAILED DESCRIPTION:
This is a Phase 1 study with 2 parts, both in healthy subjects. Part 1 is a subject- and investigator-blind, placebo-controlled, randomized, 3 period, crossover study. Part 1 will assess the safety and tolerability of LY2811376 single doses, how the body handles the drug, and the drug's effect on the body. Part 2 is a subject- and investigator-blind, placebo-controlled, randomized study to assess the safety and tolerability of a LY2811376 single dose, how the body handles the drug, and the drug's effect on the body including in cerebrospinal fluid.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and nonchild-bearing potential women
* 20 years or older
* Body mass index between 18-32kg/m2

Exclusion Criteria:

* Taking over-the-counter or prescription medication with the exception of vitamins or minerals or stable doses of thyroid or estrogen hormone replacement.
* Smoke more than 10 cigarettes per day.
* Consume more than 5 cups of coffee per day.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2008-12; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Clinical Effects | Predose and up to Day 6 of each period

SECONDARY OUTCOMES:
Plasma concentration of LY2811376 (Cmax) | Predose and up to Day 6 of each period
Plasma concentration of LY2811376 (AUC) | Predose and up to Day 6 of each period
Amyloid beta 1-40 plasma concentrations | Predose and up to Day 6 of each period
Cerebrospinal fluid (CSF) concentration of LY2811376 (Cmax) (Part 2 only) | Predose and up to 36 hours
Cerebrospinal fluid (CSF) concentration of LY2811376 (AUC) (Part 2 only) | Predose and up to 36 hours
Amyloid beta 1-40 cerebrospinal fluid CSF concentrations (Part 2 only) | Predose and up to 36 hours

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Glendale, California, United States

REFERENCES:
- [Derived] Portelius E, Dean RA, Andreasson U, Mattsson N, Westerlund A, Olsson M, Demattos RB, Racke MM, Zetterberg H, May PC, Blennow K. beta-site amyloid precursor protein-cleaving enzyme 1(BACE1) inhibitor treatment induces Abeta5-X peptides through alternative amyloid precursor protein cleavage. Alzheimers Res Ther. 2014 Nov 17;6(5-8):75. doi: 10.1186/s13195-014-0075-0. eCollection 2014. PMID 25404952